CLINICAL TRIAL: NCT00547937
Title: Nitrate and Oxidative Stress in Sleep Apnea Syndrome. Effect of Continuous Positive Airway Pressure
Brief Title: Sleep Apnea and Oxidative Stress and Nitric Oxide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: NO-OE-SAHS
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-10

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep Apnea; Oxidative Stress; Nitric oxide; Cardiovascular disease
MeSH Terms: conditions — Sleep Apnea Syndromes; Cardiovascular Diseases | interventions — Continuous Positive Airway Pressure; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham-CPAP (Sham Comparator): The sham CPAP device consisted of a conventional CPAP device, in which the area of the exhalation port was amplified, thereby nearly cancelling nasal pressure; an orifice resistor was connected between the tubing and the CPAP unit that loads the blower with the same airflow resistance as in effective CPAP
  Interventions: Device: nasal continuous positive airway pressure (CPAP) therapy
- CPAP (Active Comparator)
  Interventions: Device: nasal continuous positive airway pressure (CPAP) therapy

INTERVENTIONS:
Device: nasal continuous positive airway pressure (CPAP) therapy — Nocturnal ventilation through a nasal mask to avoid sleep apneas

SUMMARY:
Background: Previous studies present contradictory data concerning obstructive sleep apnea syndrome (OSAS), lipid oxidation and nitric oxide (NO) bioavailability. This study was aimed: (1) to compare the concentration of 8-isoprostane and total nitrate and nitrite (NOx) in plasma of middle aged males with OSAS and no other known comorbidity and carefully matched healthy controls of the same age and gender; and (2) to test the hypothesis that nasal continuous positive airway pressure (CPAP) therapy, might attenuate oxidative stress and nitrate deficiency.

DETAILED DESCRIPTION:
We performed a single-center, prospective, randomized, double-blind, placebo-controlled and cross-over clinical study, in which patients received CPAP and sham therapy for two 12-week periods. Baseline measurements in healthy controls matched for age and gender were also obtained. At recruitment, 24-h blood pressure monitoring (ABPM), an echocardiogram (to rule out any cardiac dysfunction) and a sleep study was obtained in all participants . After fasting overnight, a venous blood sample (anti-coagulated with dipotassium EDTA, for 8-isoprostane and total nitrate and nitrite concentration (NOx) determinations) and a urine sample were collected in all of them between 08:00 and 10:00 hours. Within 30 minutes of blood collection, plasma was obtained by centrifugation at 3000 rpm for 15 min. All plasma samples were stored at -60°C until analysis. Patients with OSAS underwent a full-night CPAP titration study using an automated pressure setting device (Auto Set; ResMed, Sydney, Australia). Compliance with therapy was obtained from a built-in run-time counter. After 12 weeks, CPAP device was switched to the alternate mode of therapy and ABPM,, plasma and urine sampling were repeated in patients

ELIGIBILITY:
Inclusion Criteria:

* apnea-hypopnea index (AHI) ≥10 h-1
* excessive daytime sleepiness defined by an Epworth scale score ≥11 points
* no treatment for OSAS. Inclusion criteria for healthy control subjects were AHI <5 h-1 and Epworth sleepiness scale <10.

Exclusion Criteria:

* unwillingness or inability to participate in the study
* obstructive or restrictive lung disease as identified by pulmonary function testing
* use of cardioactive drugs
* cardiac rhythm disturbances, including sinus bradycardia and sinus tachycardia
* known arterial hypertension, or 24-hour mean blood pressure of 135 and/or 85 mm Hg or more
* left ventricular ejection fraction <50%, ischemic or valve heart disease, hypertrophic, restrictive or infiltrative cardiomyopathy, pericardial disease or stroke, by history, physical examination, ECG, chest radiography, conventional exercise stress testing, and echocardiography
* diabetes mellitus, by history or 2 random blood glucose levels ≥126 mg/dl
* morbid obesity (body mass index >40 Kg/m2)
* daytime hypoxemia (PaO2 <70 mm Hg) or hypercapnia (PaCO2 >45 mm Hg)
* need to change medication
* hospital admission for 10 or more days
* average nightly CPAP usage less than 3.5 hours.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-05; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
concentration of 8-isoprostane and total nitrate and nitrite (NOx) in plasma | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Alonso, MD, Principal Investigator — Sociedad Española de Neumología y Cirugía Torácica
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain